CLINICAL TRIAL: NCT02932904
Title: A Randomized, Double-Blind, Parallel Group, Placebo- and Active-Controlled, Phase 4 Study Evaluating the Effect of Vortioxetine 10 and 20 mg/Day vs Paroxetine 20 mg/Day on Sexual Functioning in Healthy Subjects
Brief Title: Effect of Vortioxetine, Paroxetine, and Placebo on Sexual Functioning in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vortioxetine-4001; U1111-1174-1779 (Other: WHO)
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — Vortioxetine; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg, overencapsulated tablets, orally, once daily for up to 5 weeks.
  Interventions: Drug: Vortioxetine
- Vortioxetine 20 mg (Experimental): Vortioxetine 10 mg, overencapsulated tablets, orally, once daily for up to 1 week followed by vortioxetine 20 mg, overencapsulated tablets, orally, once daily from Week 2, up to 4 weeks.
  Interventions: Drug: Vortioxetine
- Paroxetine 20 mg (Active Comparator): Paroxetine 20 mg, overencapsulated tablets, orally, once daily for up to 5 weeks.
  Interventions: Drug: Paroxetine
- Placebo (Placebo Comparator): Vortioxetine placebo matching-capsules, orally, once daily for up to 5 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine Overencapsulated Tablet
  Arms: Vortioxetine 10 mg; Vortioxetine 20 mg
Drug: Paroxetine — Paroxetine Overencapsulated Tablets.
  Arms: Paroxetine 20 mg
Drug: Placebo — Vortioxetine Placebo-matching Capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of vortioxetine (10 and 20 mg, once daily) versus paroxetine (20 mg, once daily) on sexual functioning in healthy participants after 5 weeks of double-blind treatment.

DETAILED DESCRIPTION:
The drug being tested in this study is called vortioxetine. This study will look at the effect of treatment on sexual functioning in healthy participants.

The study will enroll approximately 352 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the four treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Vortioxetine 10 mg
* Vortioxetine 20 mg
* Paroxetine 20 mg
* Placebo (dummy inactive pill) - this is a capsule that looks like the study drug but has no active ingredient

All participants will be asked to take one tablet/capsule, daily, orally for up to 5 weeks.

This multicenter trial will be conducted in United States. The overall time to participate in this study is approximately 7 weeks. Participants will be contacted by telephone 2 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is sexually active and has been in a steady relationship and plans to remain in that relationship for the duration of the study.
2. Has a body mass index (BMI) of 18 to 35 kg/m^2, inclusive, at the Screening and Baseline Visits.
3. If female, has a regular menstrual cycle.
4. Has normal sexual functioning, as defined by a Changes in Sexual Functioning Questionnaire (CSFQ-14) total score >47 (men) or >41 (women) at the Screening and Baseline Visits.
5. If females, taking allowed hormonal contraceptives is on a stable dose for ≥3 months prior to the Baseline Visit and continues on the stable dose for the duration of the study.

Exclusion Criteria:

1. Has received vortioxetine and/or paroxetine in a previous clinical study or as a therapeutic agent.
2. Is positive for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, or human immunodeficiency virus (HIV) at the Screening Visit or has any known sexually transmitted diseases.
3. Has glycosylated hemoglobin (HbA1c) ≥7% at the Screening Visit.
4. Has a clinically significant abnormal electrocardiogram (ECG) at the Screening Visit.
5. Has a known history of or currently has increased intraocular pressure or is at risk of acute narrow-angle glaucoma.
6. Has a history of depression or any other psychiatric illness.
7. Has a significant risk of suicide according to the investigator's clinical judgment, or has made a suicide attempt in the previous 6 months.
8. Has current sexual dysfunction, or a history of a diagnosis or treatment of sexual dysfunction.
9. Has had a surgical or medical procedure on reproductive/genitourinary organs (excluding uncomplicated vasectomy and tubal ligation).
10. If female, has polycystic ovarian syndrome.
11. Has hypogonadism or has a free testosterone value outside the normal range at the Screening Visit that is indicative of hypogonadism.
12. Has a thyroid-stimulating hormone (TSH) value outside the normal range at the Screening Visit that is deemed clinically significant by the investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 361 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (15):
- United States (15):
  - Encino, California
  - Long Beach, California
  - Torrance, California
  - Jacksonville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Portland, Oregon
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 16 investigative sites in the United States from 21 November 2016 to 09 June 2017.
Pre-assignment Details: Healthy volunteers were randomized in a 1:1:1:1 ratio to one of 4 treatment arms: vortioxetine 10 mg, vortioxetine 20 mg, paroxetine or placebo.
Period: Overall Study
Arm/Group | Placebo | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Started | 92 | 85 | 91 | 93
Treated | 91 | 84 | 91 | 91
Completed | 76 | 67 | 68 | 79
Not Completed | 16 | 18 | 23 | 14
Not completed — Reason not Specified | 1 | 0 | 2 | 2
Not completed — Noncompliance with Study Drug | 2 | 3 | 3 | 4
Not completed — Pregnancy | 0 | 1 | 1 | 0
Not completed — Study Termination | 0 | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 2 | 1 | 4 | 2
Not completed — Lost to Follow-up | 5 | 3 | 6 | 0
Not completed — Significant Protocol Deviation | 2 | 3 | 6 | 1
Not completed — Pretreatment Event/Adverse Event | 3 | 5 | 1 | 3
Not completed — Randomized But Not Treated | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg | Total
Number analyzed (Participants) | 92 | 85 | 91 | 93 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All randomized participants.
  years | 27.8 (5.45) | 28.9 (5.96) | 28.1 (5.56) | 28.8 (5.91) | 28.4 (5.72)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All randomized participants.
  Participants
    Female | 46 | 42 | 44 | 44 | 176
    Male | 46 | 43 | 47 | 49 | 185
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: All randomized participants.
  Participants
    Hispanic or Latino | 21 | 20 | 25 | 18 | 84
    Non-Hispanic and Latino | 71 | 65 | 66 | 75 | 277
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: All randomized participants.
  Participants
    American Indian or Alaska Native | 0 | 0 | 3 | 0 | 3
    Asian | 7 | 3 | 2 | 3 | 15
    Black or African American | 30 | 29 | 31 | 34 | 124
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
    White | 51 | 49 | 52 | 55 | 207
    Multiracial | 4 | 3 | 3 | 1 | 11
Region of Enrollment [Count of Participants; unit: Participants] — Population: All randomized participants.
  Participants
    United States | 92 | 85 | 91 | 93 | 361
Median Age Categories [Count of Participants; unit: Participants] — Population: All randomized participants.
  Participants
    ≤ 28 Years | 51 | 43 | 52 | 47 | 193
    > 28 Years | 41 | 42 | 39 | 46 | 168
Race Categories [Count of Participants; unit: Participants] — Population: All randomized participants.
  Participants
    White | 51 | 49 | 52 | 55 | 207
    Non-white | 41 | 36 | 39 | 38 | 154
Height [Mean (Standard Deviation); unit: cm] — Population: All randomized participants.
  cm | 172.0 (10.75) | 172.1 (10.59) | 171.3 (9.14) | 170.8 (10.04) | 171.5 (10.12)
Weight [Mean (Standard Deviation); unit: kg] — Population: All randomized participants.
  kg | 76.49 (15.523) | 80.19 (16.808) | 78.67 (14.850) | 75.12 (13.282) | 77.56 (15.192)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: All randomized participants.
  kg/m^2 | 25.72 (3.925) | 26.91 (4.245) | 26.77 (4.306) | 25.70 (3.668) | 26.26 (4.062)
Smoking Classification [Count of Participants; unit: Participants] — Population: All randomized participants.
  Participants
    Participant has never smoked | 73 | 70 | 70 | 77 | 290
    Participant is a current smoker | 7 | 2 | 4 | 7 | 20
    Participant is an ex-smoker | 12 | 13 | 17 | 9 | 51
Female Reproductive Status [Count of Participants; unit: Participants] — Population: All randomized participants.
  Participants
    Surgically sterile | 3 | 4 | 2 | 3 | 12
    Female of childbearing potential | 43 | 38 | 42 | 41 | 164
    NA/Participant is male | 46 | 43 | 47 | 49 | 185
Duration of Menstruation [Mean (Standard Deviation); unit: days] — Population: All randomized participants. Here, n=number analysed is the female participants who were evaluable for this parameter at baseline.
  days
    number analyzed (Participants) | 45 | 42 | 44 | 43 | 174
    (all) | 4.9 (1.36) | 4.4 (1.27) | 4.2 (1.27) | 4.6 (1.37) | 4.5 (1.33)
Duration of Menstrual Cycle [Mean (Standard Deviation); unit: days] — Population: All randomized participants. Here, n=number analysed is the female participants who were evaluable for this parameter at baseline.
  days
    number analyzed (Participants) | 45 | 42 | 44 | 43 | 174
    (all) | 28.9 (5.35) | 28.3 (2.56) | 28.2 (7.07) | 28.0 (6.94) | 28.4 (5.75)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Changes in Sexual Functioning Questionnaire (CSFQ-14) Total Score Difference for Vortioxetine Versus Paroxetine at Week 5 in Full Analysis Set (FAS)
Description: The CSFQ-14 is a structured, self-reported questionnaire designed to measure illness- and medication-related changes in sexual functioning consisting of 14 items that measure sexual functioning as a total score (14 items) and on the subscales of pleasure (1 item), desire/frequency (2 items), desire/interest (3 items), arousal (3 items), orgasm (3 items) and 2 additional items are included in the total score, but do not map to a specific phase of the sexual response cycle, rated on a 5-point scale from 1 to 5 with a total score range from 14 to 70. Higher scores reflect higher sexual functioning. A negative change from baseline indicates that symptoms have worsened.
Time Frame: Baseline and Week 5
Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid postbaseline value for assessment of primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 83 | 85 | 91
score on a scale
  Baseline | 59.27 (0.584) | 58.56 (0.578) | 59.43 (0.560)
  Change from Baseline at Week 5 | -3.56 (0.758) | -0.82 (0.752) | -2.51 (0.727)
Statistical Analysis 1: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; ANCOVA with last observation carried forward (LOCF) model was used for p-value with treatment, pooled center, and gender as fixed factors and with baseline CSFQ-14 total score as a covariate; Test type: Superiority; p = 0.009, ANCOVA with LOCF — The comparisons were between each vortioxetine dose (10 or 20 mg) and paroxetine, and the Holm-Bonferroni method was used to adjust for multiplicity and control the familywise type I error rate at a significance level of 0.05; Least square (LS) Mean Difference = 2.74, 95% CI 2-sided [0.69 to 4.78], Standard Error of Mean 1.040
Statistical Analysis 2: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; ANCOVA model with the LOCF method was used for p-value with treatment, pooled center, and gender as fixed factors and with baseline CSFQ-14 total score as a covariate; Test type: Superiority; p = 0.303, ANCOVA with LOCF — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 1.05, 95% CI 2-sided [-0.95 to 3.05], Standard Error of Mean 1.017

2. Secondary Outcome: Change From Baseline in the CSFQ-14 Total Score Difference for Vortioxetine Versus Paroxetine at Weeks 1, 2, 3 and 4
Description: as for outcome 1
Time Frame: Baseline and Weeks 1, 2, 3 and 4
Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid postbaseline value for assessment of primary endpoint. Here, number analyzed are the participants who were evaluated for this outcome measure in the FAS.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 83 | 85 | 91
score on a scale
  Week 1: number analyzed (Participants) | 82 | 84 | 91
  Week 1 | -1.67 (0.457) | -0.54 (0.453) | -0.38 (0.436)
  Week 2 | -2.40 (0.617) | -1.18 (0.612) | -1.55 (0.592)
  Week 3 | -2.77 (0.661) | -0.77 (0.655) | -2.36 (0.633)
  Week 4 | -3.11 (0.688) | -1.20 (0.683) | -2.43 (0.659)
Statistical Analysis 1: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; Week 1, ANCOVA model with the LOCF method was used for p-value with treatment, pooled center, and gender as fixed factors and with baseline CSFQ-14 total score as a covariate; Test type: Superiority; p = 0.072, ANCOVA with LOCF; LS Mean Difference = 1.13, 95% CI 2-sided [-0.10 to 2.37], Standard Error of Mean 0.627
Statistical Analysis 2: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.035, ANCOVA with LOCF; LS Mean Difference = 1.29, 95% CI 2-sided [0.09 to 2.50], Standard Error of Mean 0.612
Statistical Analysis 3: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; Week 2, ANCOVA model with the LOCF method was used for p-value with treatment, pooled center, and gender as fixed factors and with baseline CSFQ-14 total score as a covariate; Test type: Superiority; p = 0.149, ANCOVA with LOCF; LS Mean Difference = 1.22, 95% CI 2-sided [-0.44 to 2.89], Standard Error of Mean 0.846
Statistical Analysis 4: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.303, ANCOVA with LOCF; LS Mean Difference = 0.85, 95% CI 2-sided [-0.78 to 2.48], Standard Error of Mean 0.828
Statistical Analysis 5: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; Week 3, ANCOVA model with the LOCF method was used for p-value with treatment, pooled center, and gender as fixed factors and with baseline CSFQ-14 total score as a covariate; Test type: Superiority; p = 0.028, ANCOVA with LOCF; LS Mean Difference = 2.00, 95% CI 2-sided [0.22 to 3.78], Standard Error of Mean 0.906
Statistical Analysis 6: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.645, ANCOVA with LOCF; LS Mean Difference = 0.41, 95% CI 2-sided [-1.33 to 2.15], Standard Error of Mean 0.886
Statistical Analysis 7: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; Week 4, ANCOVA model with the LOCF method was used for p-value with treatment, pooled center, and gender as fixed factors and with baseline CSFQ-14 total score as a covariate; Test type: Superiority; p = 0.043, ANCOVA with LOCF; LS Mean Difference = 1.91, 95% CI 2-sided [0.06 to 3.77], Standard Error of Mean 0.943
Statistical Analysis 8: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.465, ANCOVA with LOCF; LS Mean Difference = 0.68, 95% CI 2-sided [-1.14 to 2.49], Standard Error of Mean 0.923

3. Secondary Outcome: Change From Baseline in CSFQ-14 Total Score Difference for Paroxetine Versus Placebo at Weeks 1, 2, 3, 4 and 5
Description: as for outcome 1
Time Frame: Baseline and Weeks 1, 2, 3, 4 and 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Paroxetine 20 mg
Number analyzed (Participants) | 89 | 83
score on a scale
  Week 1: number analyzed (Participants) | 89 | 82
  Week 1 | -0.05 (0.440) | -1.67 (0.457)
  Week 2 | -1.11 (0.598) | -2.40 (0.617)
  Week 3 | -0.91 (0.639) | -2.77 (0.661)
  Week 4 | -0.62 (0.666) | -3.11 (0.688)
  Week 5 | -0.79 (0.734) | -3.56 (0.758)
Statistical Analysis 1: Comparison: Placebo vs Paroxetine 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.009, ANCOVA with LOCF; LS Mean Difference = -1.63, 95% CI 2-sided [-2.84 to -0.41], Standard Error of Mean 0.616
Statistical Analysis 2: Comparison: Placebo vs Paroxetine 20 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.123, ANCOVA with LOCF; LS Mean Difference = -1.29, 95% CI 2-sided [-2.93 to 0.35], Standard Error of Mean 0.834
Statistical Analysis 3: Comparison: Placebo vs Paroxetine 20 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.039, ANCOVA with LOCF; LS Mean Difference = -1.85, 95% CI 2-sided [-3.61 to -0.10], Standard Error of Mean 0.892
Statistical Analysis 4: Comparison: Placebo vs Paroxetine 20 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.008, ANCOVA with LOCF; LS Mean Difference = -2.49, 95% CI 2-sided [-4.32 to -0.66], Standard Error of Mean 0.929
Statistical Analysis 5: Comparison: Placebo vs Paroxetine 20 mg; Week 5, ANCOVA model with the LOCF method was used for p-value with treatment, pooled center, and gender as fixed factors and with baseline CSFQ-14 total score as a covariate; Test type: Superiority; p = 0.007, ANCOVA with LOCF; LS Mean Difference = -2.77, 95% CI 2-sided [-4.78 to -0.75], Standard Error of Mean 1.024

4. Secondary Outcome: Change From Baseline in CSFQ-14 Total Score Difference for Vortioxetine Versus Placebo at Weeks 1, 2, 3, 4 and 5
Description: as for outcome 1
Time Frame: Baseline and Weeks 1, 2, 3, 4 and 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 89 | 85 | 91
score on a scale
  Week 1: number analyzed (Participants) | 89 | 84 | 91
  Week 1 | -0.05 (0.440) | -0.54 (0.453) | -0.38 (0.436)
  Week 2 | -1.11 (0.598) | -1.18 (0.612) | -1.55 (0.592)
  Week 3 | -0.91 (0.639) | -0.77 (0.655) | -2.36 (0.633)
  Week 4 | -0.62 (0.666) | -1.20 (0.683) | -2.43 (0.659)
  Week 5 | -0.79 (0.734) | -0.82 (0.752) | -2.51 (0.727)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.419, ANCOVA with LOCF; LS Mean Difference = -0.50, 95% CI 2-sided [-1.70 to 0.71], Standard Error of Mean 0.612
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.581, ANCOVA with LOCF; LS Mean Difference = -0.33, 95% CI 2-sided [-1.51 to 0.85], Standard Error of Mean 0.600
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 10 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.938, ANCOVA with LOCF; LS Mean Difference = -0.06, 95% CI 2-sided [-1.69 to 1.56], Standard Error of Mean 0.828
Statistical Analysis 4: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.592, ANCOVA with LOCF; LS Mean Difference = -0.44, 95% CI 2-sided [-2.04 to 1.17], Standard Error of Mean 0.814
Statistical Analysis 5: Comparison: Placebo vs Vortioxetine 10 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.870, ANCOVA with LOCF; LS Mean Difference = 0.15, 95% CI 2-sided [-1.60 to 1.89], Standard Error of Mean 0.886
Statistical Analysis 6: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.098, ANCOVA with LOCF; LS Mean Difference = -1.44, 95% CI 2-sided [-3.16 to 0.27], Standard Error of Mean 0.871
Statistical Analysis 7: Comparison: Placebo vs Vortioxetine 10 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.532, ANCOVA with LOCF; LS Mean Difference = -0.58, 95% CI 2-sided [-2.39 to 1.24], Standard Error of Mean 0.923
Statistical Analysis 8: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.046, ANCOVA with LOCF; LS Mean Difference = -1.82, 95% CI 2-sided [-3.60 to -0.03], Standard Error of Mean 0.907
Statistical Analysis 9: Comparison: Placebo vs Vortioxetine 10 mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.977, ANCOVA with LOCF; LS Mean Difference = -0.03, 95% CI 2-sided [-2.03 to 1.97], Standard Error of Mean 1.018
Statistical Analysis 10: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.087, ANCOVA with LOCF; LS Mean Difference = -1.72, 95% CI 2-sided [-3.68 to 0.25], Standard Error of Mean 1.000

5. Secondary Outcome: Percentage of Participants Meeting Criteria for Sexual Dysfunction at Weeks 1, 2, 3, 4 and 5
Description: Sexual dysfunction is defined as CSFQ-14 score ≤47 for men and ≤41 for women.
Time Frame: Weeks 1, 2, 3, 4 and 5
Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid postbaseline value for assessment of primary endpoint. Missing values were imputed by using LOCF. Here, number analyzed are the participants who were evaluated for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 89 | 83 | 85 | 91
percentage of participants
  Week 1: number analyzed (Participants) | 89 | 82 | 84 | 91
  Week 1 | 2.2 | 2.4 | 1.2 | 1.1
  Week 2 | 7.9 | 8.4 | 3.5 | 2.2
  Week 3 | 4.5 | 8.4 | 3.5 | 6.6
  Week 4 | 4.5 | 9.6 | 4.7 | 7.7
  Week 5 | 3.4 | 9.6 | 5.9 | 9.9
Statistical Analysis 1: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; Week 1; Test type: Superiority — Odds ratio, 95% confidence intervals and p-values are from logistic regression model using the rate of subjects that shifted from normal at baseline to abnormal after baseline as the response and explanatory variables for treatment, baseline CSFQ-14 total score, and gender; p = 0.515, Regression, Logistic; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.037 to 5.201]
Statistical Analysis 2: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; Week 1; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.677, Regression, Logistic; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.049 to 7.051]
Statistical Analysis 3: Comparison: Placebo vs Paroxetine 20 mg; Week 1; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.720, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.181 to 11.912]
Statistical Analysis 4: Comparison: Placebo vs Vortioxetine 10 mg; Week 1; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.732, Regression, Logistic; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.053 to 7.861]
Statistical Analysis 5: Comparison: Placebo vs Vortioxetine 20 mg; Week 1; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.913, Regression, Logistic; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.066 to 11.303]
Statistical Analysis 6: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; Week 2; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.164, Regression, Logistic; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.090 to 1.507]
Statistical Analysis 7: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; Week 2; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.098, Regression, Logistic; Odds Ratio (OR) = 0.25, 95% CI 2-sided [0.050 to 1.287]
Statistical Analysis 8: Comparison: Placebo vs Paroxetine 20 mg; Week 2; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.758, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.383 to 3.731]
Statistical Analysis 9: Comparison: Placebo vs Vortioxetine 10 mg; Week 2; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.256, Regression, Logistic; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.107 to 1.814]
Statistical Analysis 10: Comparison: Placebo vs Vortioxetine 20 mg; Week 2; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.154, Regression, Logistic; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.059 to 1.561]
Statistical Analysis 11: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; Week 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.160, Regression, Logistic; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.087 to 1.497]
Statistical Analysis 12: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; Week 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.744, Regression, Logistic; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.252 to 2.679]
Statistical Analysis 13: Comparison: Placebo vs Paroxetine 20 mg; Week 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.194, Regression, Logistic; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.636 to 9.317]
Statistical Analysis 14: Comparison: Placebo vs Vortioxetine 10 mg; Week 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.871, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.181 to 4.261]
Statistical Analysis 15: Comparison: Placebo vs Vortioxetine 20 mg; Week 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.329, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.497 to 8.037]
Statistical Analysis 16: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; Week 4; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.187, Regression, Logistic; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.119 to 1.514]
Statistical Analysis 17: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; Week 4; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.729, Regression, Logistic; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.273 to 2.476]
Statistical Analysis 18: Comparison: Placebo vs Paroxetine 20 mg; Week 4; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.133, Regression, Logistic; Odds Ratio (OR) = 2.71, 95% CI 2-sided [0.739 to 9.917]
Statistical Analysis 19: Comparison: Placebo vs Vortioxetine 10 mg; Week 4; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.852, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.266 to 4.961]
Statistical Analysis 20: Comparison: Placebo vs Vortioxetine 20 mg; Week 4; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.240, Regression, Logistic; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.585 to 8.472]
Statistical Analysis 21: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; Week 5; Test type: Superiority — Odds ratio, 95% confidence intervals and p-values are from logistic regression model using rate of subjects that shifted from normal at baseline to abnormal after baseline as response and explanatory variables for treatment, baseline CSFQ-14 total score, and gender; p = 0.317, Regression, Logistic; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.166 to 1.789]
Statistical Analysis 22: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; Week 5; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.790, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.410 to 3.233]
Statistical Analysis 23: Comparison: Placebo vs Paroxetine 20 mg; Week 5; Test type: Superiority — [test comment as in outcome 5, analysis 21]; p = 0.073, Regression, Logistic; Odds Ratio (OR) = 3.64, 95% CI 2-sided [0.888 to 14.911]
Statistical Analysis 24: Comparison: Placebo vs Vortioxetine 10 mg; Week 5; Test type: Superiority — [test comment as in outcome 5, analysis 21]; p = 0.371, Regression, Logistic; Odds Ratio (OR) = 1.98, 95% CI 2-sided [0.442 to 8.902]
Statistical Analysis 25: Comparison: Placebo vs Vortioxetine 20 mg; Week 5; Test type: Superiority — [test comment as in outcome 5, analysis 21]; p = 0.046, Regression, Logistic; Odds Ratio (OR) = 4.19, 95% CI 2-sided [1.027 to 17.063]

6. Secondary Outcome: Change From Baseline in CSFQ-14 Subscales 5 Dimensions at Weeks 1, 2, 3, 4 and 5
Description: The CSFQ-14 is a structured, self-reported questionnaire designed to measure illness- and medication-related changes in sexual functioning consisting of 14 items that measure sexual functioning on the subscales of pleasure (1 item, score range 1-5), desire/frequency (2 items, score range 2-10), desire/interest (3 items, score range 3-15), arousal (3 items, score range 3-15), and orgasm (3 items, score range 3-15), rated on a 5-point scale from 1 to 5. Higher scores reflect higher sexual functioning. A negative change from baseline indicates that symptoms have worsened.
Time Frame: Baseline and Weeks 1, 2, 3, 4 and 5
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 89 | 83 | 85 | 91
score on a scale
  Pleasure Score: Week 1: number analyzed (Participants) | 89 | 82 | 84 | 91
  Pleasure Score: Week 1 | -0.07 (0.064) | -0.36 (0.066) | -0.13 (0.065) | -0.15 (0.063)
  Pleasure Score: Week 2 | -0.26 (0.079) | -0.38 (0.082) | -0.25 (0.081) | -0.26 (0.078)
  Pleasure Score: Week 3 | -0.23 (0.085) | -0.44 (0.088) | -0.18 (0.087) | -0.42 (0.084)
  Pleasure Score: Week 4 | -0.18 (0.085) | -0.38 (0.088) | -0.31 (0.087) | -0.37 (0.084)
  Pleasure Score: Week 5 | -0.21 (0.086) | -0.47 (0.089) | -0.16 (0.088) | -0.33 (0.085)
  Desire/Frequency Score: Week 1: number analyzed (Participants) | 89 | 82 | 84 | 91
  Desire/Frequency Score: Week 1 | -0.03 (0.097) | -0.35 (0.100) | -0.07 (0.099) | -0.23 (0.096)
  Desire/Frequency Score: Week 2 | -0.30 (0.118) | -0.46 (0.122) | -0.25 (0.120) | -0.46 (0.116)
  Desire/Frequency Score: Week 3 | -0.33 (0.128) | -0.62 (0.132) | -0.23 (0.131) | -0.50 (0.127)
  Desire/Frequency Score: Week 4 | -0.25 (0.126) | -0.55 (0.130) | -0.20 (0.129) | -0.43 (0.125)
  Desire/Frequency Score: Week 5 | -0.28 (0.141) | -0.66 (0.145) | -0.15 (0.144) | -0.49 (0.139)
  Desire/Interest Score: Week 1: number analyzed (Participants) | 89 | 82 | 84 | 91
  Desire/Interest Score: Week 1 | 0.12 (0.162) | -0.15 (0.169) | -0.16 (0.167) | 0.09 (0.161)
  Desire/Interest Score: Week 2 | -0.09 (0.181) | -0.38 (0.186) | -0.11 (0.185) | -0.22 (0.179)
  Desire/Interest Score: Week 3 | -0.16 (0.193) | -0.47 (0.200) | -0.01 (0.198) | -0.28 (0.191)
  Desire/Interest Score: Week 4 | -0.11 (0.200) | -0.52 (0.206) | -0.18 (0.204) | -0.35 (0.198)
  Desire/Interest Score: Week 5 | -0.14 (0.215) | -0.73 (0.223) | -0.05 (0.221) | -0.33 (0.213)
  Arousal/Excitement/Erection Score: Week 1: number analyzed (Participants) | 89 | 82 | 84 | 91
  Arousal/Excitement/Erection Score: Week 1 | -0.01 (0.136) | -0.30 (0.141) | -0.05 (0.140) | -0.03 (0.135)
  Arousal/Excitement/Erection Score: Week 2 | -0.34 (0.175) | -0.47 (0.181) | -0.35 (0.179) | -0.30 (0.174)
  Arousal/Excitement/Erection Score: Week 3 | -0.22 (0.182) | -0.43 (0.188) | -0.08 (0.186) | -0.51 (0.180)
  Arousal/Excitement/Erection Score: Week 4 | -0.11 (0.181) | -0.54 (0.187) | -0.10 (0.185) | -0.54 (0.179)
  Arousal/Excitement/Erection Score: Week 5 | -0.19 (0.195) | -0.67 (0.202) | -0.03 (0.200) | -0.54 (0.193)
  Orgasm/Completion/Ejaculation Score: Week 1: number analyzed (Participants) | 89 | 82 | 84 | 91
  Orgasm/Completion/Ejaculation Score: Week 1 | -0.12 (0.130) | -0.48 (0.135) | -0.22 (0.134) | -0.15 (0.129)
  Orgasm/Completion/Ejaculation Score: Week 2 | -0.21 (0.158) | -0.61 (0.164) | -0.26 (0.162) | -0.37 (0.157)
  Orgasm/Completion/Ejaculation Score: Week 3 | -0.20 (0.176) | -0.75 (0.183) | -0.33 (0.180) | -0.67 (0.175)
  Orgasm/Completion/Ejaculation Score: Week 4 | -0.14 (0.194) | -1.04 (0.201) | -0.45 (0.199) | -0.72 (0.192)
  Orgasm/Completion/Ejaculation Score: Week 5 | -0.12 (0.206) | -1.09 (0.214) | -0.42 (0.211) | -0.79 (0.204)

7. Secondary Outcome: Change From Baseline in CSFQ-14 3 Phases of the Sexual Response Cycle (Desire, Arousal, and Orgasm/Completion) at Weeks 1, 2, 3, 4 and 5
Description: The CSFQ-14 is a structured, self-reported questionnaire designed to measure illness- and medication-related changes in sexual functioning consisting of 14 items that measure sexual functioning on the 3 phases of the sexual response cycle , desire (5 items, score range 5-25), arousal (3 items, score range 3-15), and orgasm (3 items, score range 3-15), rated on a 5-point scale from 1 to 5. Higher scores reflect higher sexual functioning. A negative change from baseline indicates that symptoms have worsened.
Time Frame: Baseline and Weeks 1, 2, 3, 4 and 5
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 89 | 83 | 85 | 91
score on a scale
  Desire Score: Week 1: number analyzed (Participants) | 89 | 82 | 84 | 91
  Desire Score: Week 1 | 0.09 (0.225) | -0.50 (0.234) | -0.23 (0.232) | -0.14 (0.223)
  Desire Score: Week 2 | -0.40 (0.260) | -0.83 (0.269) | -0.34 (0.266) | -0.68 (0.258)
  Desire Score: Week 3 | -0.50 (0.286) | -1.09 (0.296) | -0.22 (0.293) | -0.77 (0.284)
  Desire Score: Week 4 | -0.36 (0.297) | -1.07 (0.307) | -0.37 (0.304) | -0.77 (0.294)
  Desire Score: Week 5 | -0.42 (0.325) | -1.38 (0.336) | -0.19 (0.333) | -0.82 (0.322)
  Arousal Score: Week 1: number analyzed (Participants) | 89 | 82 | 84 | 91
  Arousal Score: Week 1 | -0.01 (0.136) | -0.30 (0.141) | -0.05 (0.140) | -0.03 (0.135)
  Arousal Score: Week 2 | -0.34 (0.175) | -0.47 (0.181) | -0.35 (0.179) | -0.30 (0.174)
  Arousal Score: Week 3 | -0.22 (0.182) | -0.43 (0.188) | -0.08 (0.186) | -0.51 (0.180)
  Arousal Score: Week 4 | -0.11 (0.181) | -0.54 (0.187) | -0.10 (0.185) | -0.54 (0.179)
  Arousal Score: Week 5 | -0.19 (0.195) | -0.67 (0.202) | -0.03 (0.200) | -0.54 (0.193)
  Orgasm/Completion/Ejaculation Score: Week 1: number analyzed (Participants) | 89 | 82 | 84 | 91
  Orgasm/Completion/Ejaculation Score: Week 1 | -0.12 (0.130) | -0.48 (0.135) | -0.22 (0.134) | -0.15 (0.129)
  Orgasm/Completion/Ejaculation Score: Week 2 | -0.21 (0.158) | -0.61 (0.164) | -0.26 (0.162) | -0.37 (0.157)
  Orgasm/Completion/Ejaculation Score: Week 3 | -0.20 (0.176) | -0.75 (0.183) | -0.33 (0.180) | -0.67 (0.175)
  Orgasm/Completion/Ejaculation Score: Week 4 | -0.14 (0.194) | -1.04 (0.201) | -0.45 (0.199) | -0.72 (0.192)
  Orgasm/Completion/Ejaculation Score: Week 5 | -0.12 (0.206) | -1.09 (0.214) | -0.42 (0.211) | -0.79 (0.204)

8. Primary Outcome: Change From Baseline in the CSFQ-14 Total Score Difference for Vortioxetine Versus Paroxetine at Week 5 in Modified Full Analysis Set 1 (mFAS1)
Description: as for outcome 1
Time Frame: Baseline and Week 5
Population: mFAS1 included all participants in the FAS except those who had active drug concentrations below the limit of quantification (BLOQ) at all study visits where pharmacokinetic (PK) samples were collected.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 74 | 82 | 84
score on a scale
  Baseline | 59.13 (0.614) | 58.55 (0.582) | 59.36 (0.576)
  Change from Baseline at Week 5 | -4.01 (0.803) | -0.63 (0.763) | -2.38 (0.754)
Statistical Analysis 1: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.002, ANCOVA with LOCF — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 3.38, 95% CI 2-sided [1.25 to 5.51], Standard Error of Mean 1.082
Statistical Analysis 2: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.129, ANCOVA with LOCF — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 1.63, 95% CI 2-sided [-0.47 to 3.73], Standard Error of Mean 1.068

9. Primary Outcome: Change From Baseline in the CSFQ-14 Total Score Difference for Vortioxetine Versus Paroxetine at Week 5 in Modified Full Analysis Set 2 (mFAS2)
Description: as for outcome 1
Time Frame: Baseline and Week 5
Population: mFAS2 included all participants in the FAS except those who had drug concentrations BLOQ at any study visit where PK samples were collected.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 60 | 79 | 79
score on a scale
  Baseline | 58.73 (0.675) | 58.53 (0.589) | 59.23 (0.591)
  Change from Baseline at Week 5 | -4.78 (0.828) | -0.47 (0.724) | -1.72 (0.724)
Statistical Analysis 1: Comparison: Paroxetine 20 mg vs Vortioxetine 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA with LOCF — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 4.31, 95% CI 2-sided [2.19 to 6.43], Standard Error of Mean 1.078
Statistical Analysis 2: Comparison: Paroxetine 20 mg vs Vortioxetine 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.005, ANCOVA with LOCF — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 3.06, 95% CI 2-sided [0.95 to 5.17], Standard Error of Mean 1.072

ADVERSE EVENTS:
Time Frame: From the first dose of study drug on Day 1 until the Follow-up Contact at Week 7
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Paroxetine 20 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/84 | 0/91 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/84 | 0/91 | 0/91
Other Adverse Events (participants affected / at risk) | 36/91 | 59/84 | 52/91 | 40/91
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | Paroxetine 20 mg (N=84) | Vortioxetine 10 mg (N=91) | Vortioxetine 20 mg (N=91)
Nausea (Gastrointestinal disorders) | 4 | 22 | 26 | 18
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 1 | 3
Fatigue (General disorders) | 2 | 5 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 4 | 4
Viral upper respiratory tract infection (Infections and infestations) | 5 | 4 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 6 | 4 | 1
Somnolence (Nervous system disorders) | 4 | 10 | 7 | 7
Headache (Nervous system disorders) | 6 | 6 | 2 | 6
Dizziness (Nervous system disorders) | 1 | 6 | 0 | 1
Libido decreased (Psychiatric disorders) | 11 | 18 | 14 | 10
Orgasm abnormal (Psychiatric disorders) | 2 | 14 | 7 | 3
Anxiety (Psychiatric disorders) | 1 | 6 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 6 | 1 | 1
Ejaculation delayed (Reproductive system and breast disorders) | 0 | 5 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT02932904/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT02932904/SAP_001.pdf